CLINICAL TRIAL: NCT01873950
Title: A Double-Blind, Randomized, Placebo-Controlled Single-Dose, Five Period Crossover Study of the Electrocardiographic Effects of Ranolazine, Dofetilide, Verapamil, and Quinidine in Healthy Subjects
Brief Title: Study of the Electrocardiographic Effects of Ranolazine, Dofetilide, Verapamil, and Quinidine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: Spaulding Clinical Research LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13-011D; SCR-002
Record Dates: First submitted 2013-05-22; First posted 2013-06-10 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Drug-induced Surface ECG Changes
MeSH Terms: interventions — Ranolazine; dofetilide; Verapamil; Quinidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ranolazine 1500mg (Experimental): Ranolazine
  Interventions: Drug: Ranolazine
- Dofetilide 500mcg (Experimental): Dofetilide
  Interventions: Drug: Dofetilide
- Verapamil HCl 120 mg (Experimental): Verapamil
  Interventions: Drug: Verapamil
- Quinidine sulfate 400mg (Experimental): Quinidine sulfate
  Interventions: Drug: Quinidine sulfate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine
  Arms: Ranolazine 1500mg
Drug: Dofetilide
  Arms: Dofetilide 500mcg
Drug: Verapamil
  Arms: Verapamil HCl 120 mg
Drug: Quinidine sulfate
  Arms: Quinidine sulfate 400mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study seeks to compare 4 known QT prolonging drugs versus placebo to determine their effects on electrophysiological and other clinical parameters. The underlying purpose is to determine if depolarization and repolarization effects caused by drugs with differing ionic channel mechanisms can be distinguished from one another, and to gauge the sensitivity and specificity of novel signal analyses for detection of depolarization and repolarization changes. Secondarily, to evaluate the exposure response relationship and drug induced effects on the heart rate biomarker relationship.

DETAILED DESCRIPTION:
This will be a randomized, double blind, 5 way crossover research study in healthy male and female subjects, 18 to 35 years of age, to compare 4 known QT prolonging drugs versus placebo to determine their effects on electrophysiological and other clinical parameters. To maintain the study blind, subjects will be blindfolded during study drug administration. The cardiologists at the central ECG laboratory (Spaulding Clinical Research, LLC) will be blinded to treatment, time, and study day/subject identifiers.

Subjects who meet all of the following inclusion criteria will be eligible to participate in the study:

1. Subject signs an Institutional Review Board (IRB) approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization for sites in the United States) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 35 years of age, inclusive, who weighs at least 50 kg (110 pounds) and has a body mass index of 18 to 27 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead ECG results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Female subjects must be at least 2 years postmenopausal, surgically sterile or practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique), and not pregnant or lactating before enrollment in the study.
5. Male or female subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.
6. Subject is highly likely (as determined by the investigator) to comply with the protocol-defined procedures and to complete the study.

ELIGIBILITY:
Inclusion Criteria: Subjects who meet all of the following inclusion criteria will be eligible to participate in the study:

1. Subject signs an IRB approved written informed consent and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization for sites in the United States) before any study related procedures are performed.
2. Subject is a healthy man or woman, 18 to 35 years of age, inclusive, who weighs at least 50 kg (110 pounds) and has a body mass index of 18 to 27 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12 lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Female subjects must be at least 2 years postmenopausal, surgically sterile or practicing 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique), and not pregnant or lactating before enrollment in the study.
5. Male or female subjects must agree to practice 2 highly effective methods of birth control (as determined by the investigator or designee; one of the methods must be a barrier technique) from Screening until 30 days after the last dose of study drug.
6. Subject is highly likely (as determined by the investigator) to comply with the protocol defined procedures and to complete the study.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria will not be eligible to participate in the study:

  1. Subject has a 12 lead safety ECG result at Screening or Check in of Period 1 with evidence of any of the following abnormalities:

     * QTc using Fridericia correction (QTcF) >450 milliseconds (ms) for men and >470 ms for women
     * PR interval >220 ms
     * QRS duration >110 ms
     * Second- or third-degree atrioventricular block
     * Complete left or right bundle branch block or incomplete right bundle branch block
     * Heart rate <40 or >90 beats per minute
     * Pathological Q-waves (defined as Q wave >40 ms)
     * Ventricular pre-excitation
  2. Subject has more than 12 to 20 ectopic beats during the 3 hour Holter ECG at Screening.
  3. Subject has a history of unexplained syncope, structural heart disease, long QT syndrome, heart failure, myocardial infarction, angina, unexplained cardiac arrhythmia, torsades de pointes, ventricular tachycardia, or placement of a pacemaker or implantable defibrillator. Subjects will also be excluded if there is a family history of long QT syndrome (genetically proven or suggested by sudden death of a close relative due to cardiac causes at a young age) or Brugada syndrome.
  4. Subject has a history or current evidence of any clinically significant (as determined by the investigator) cardiovascular, dermatologic, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurologic, psychiatric, pulmonary, renal, urologic, and/or other major disease or malignancy (excluding nonmelanoma skin cancer). The investigator may allow exceptions to these criteria (e.g., stable mild joint disease [that will not interfere with or influence the leg raises/exercises required by the protocol, in the opinion of the investigator], cholecystectomy, childhood asthma) following discussion with the medical monitor.
  5. Subject has a history of thoracic surgery.
  6. Subject has any condition possibly affecting study drug absorption (e.g., gastrectomy, Crohn's disease, irritable bowel syndrome).
  7. Subject has a skin condition likely to compromise ECG electrode placement.
  8. Subject is a female with breast implants.
  9. Subject's laboratory test results at Screening or Check in of Period 1 are outside the reference ranges provided by the clinical laboratory and considered clinically significant (as determined and documented by the investigator or designee).
  10. Subject's laboratory test results at Screening or Check in of Period 1 indicate hypokalemia, hypocalcemia, or hypomagnesemia according to lower limits of the reference ranges provided by the clinical laboratory.
  11. Subject's laboratory test results at Screening or Check in of Period 1 are >2 × the upper limit of normal (ULN) for alanine aminotransferase or aspartate aminotransferase, >1.5 × ULN for bilirubin, or >1.5 × ULN for creatinine.
  12. Subject has a positive test result at Screening for human immunodeficiency virus antibody, hepatitis C antibodies, or hepatitis B surface antigen.
  13. Subject has a mean systolic blood pressure <90 or >140 mmHg or a mean diastolic blood pressure <50 or >90 mmHg at either Screening or Check in of Period 1. Blood pressure will be measured in triplicate after the subject has been resting in a supine position for a minimum of 5 minutes.
  14. Subject has a known hypersensitivity to ranolazine, dofetilide, verapamil, or quinidine or related compounds.
  15. Subject has consumed alcohol, xanthine containing products (e.g., tea, coffee, chocolate, cola), caffeine, grapefruit, or grapefruit juice within 48 hours before dosing or anticipates an inability to abstain from these products throughout the duration of the study.
  16. Subject has used nicotine containing products (e.g., cigarettes, cigars, chewing tobacco, snuff) within 6 weeks before Screening (self reported).
  17. Subject is unable to tolerate a controlled, quiet study conduct environment, including avoidance of music, television, movies, games, and activities that may cause excitement, emotional tension, or arousal during the prespecified time points (e.g., before and during ECG extraction windows).
  18. Subject is unwilling to comply with study rules, including the study specific diet, attempting to void at specified times (e.g., before ECG extraction windows), remaining quiet, awake, undistracted, motionless, and supine during specified times, and avoiding vigorous exercise as directed.
  19. Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months before Screening, has a history of alcoholism or drug/chemical/substance abuse within 2 years before Screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor), or has a positive test result for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates) at Screening or Check in of each period.
  20. Subject has used any prescription or nonprescription drugs within 14 days or 5 half lives (whichever is longer), or complementary and alternative medicines within 28 days before the first dose of study drug (excluding oral contraceptives, hormone replacement therapy, aspirin, ibuprofen, and acetaminophen).
  21. Subject is currently participating in another clinical study of an investigational drug or has been treated with any investigational drug within 30 days or 5 half lives (whichever is longer) of the compound.
  22. Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days before Check in of Period 1.
  23. Subject has any other condition that precludes his or her participation in the study (as determined by the investigator).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Sanabria, MD, Principal Investigator — Spaulding Clinical Research LLC

REFERENCES:
- [Result] Johannesen L, Vicente J, Mason JW, Sanabria C, Waite-Labott K, Hong M, Guo P, Lin J, Sorensen JS, Galeotti L, Florian J, Ugander M, Stockbridge N, Strauss DG. Differentiating drug-induced multichannel block on the electrocardiogram: randomized study of dofetilide, quinidine, ranolazine, and verapamil. Clin Pharmacol Ther. 2014 Nov;96(5):549-58. doi: 10.1038/clpt.2014.155. Epub 2014 Jul 23. PMID 25054430
- [Result] Vicente J, Johannesen L, Mason JW, Crumb WJ, Pueyo E, Stockbridge N, Strauss DG. Comprehensive T wave morphology assessment in a randomized clinical study of dofetilide, quinidine, ranolazine, and verapamil. J Am Heart Assoc. 2015 Apr 13;4(4):e001615. doi: 10.1161/JAHA.114.001615. PMID 25870186
- [Result] Vicente J, Johannesen L, Mason JW, Pueyo E, Stockbridge N, Strauss DG. Sex differences in drug-induced changes in ventricular repolarization. J Electrocardiol. 2015 Nov-Dec;48(6):1081-7. doi: 10.1016/j.jelectrocard.2015.08.004. Epub 2015 Aug 4. PMID 26324176
- [Derived] Strauss DG, Vicente J, Johannesen L, Blinova K, Mason JW, Weeke P, Behr ER, Roden DM, Woosley R, Kosova G, Rosenberg MA, Newton-Cheh C. Common Genetic Variant Risk Score Is Associated With Drug-Induced QT Prolongation and Torsade de Pointes Risk: A Pilot Study. Circulation. 2017 Apr 4;135(14):1300-1310. doi: 10.1161/CIRCULATIONAHA.116.023980. Epub 2017 Feb 17. PMID 28213480
- [Derived] Vicente J, Johannesen L, Hosseini M, Mason JW, Sager PT, Pueyo E, Strauss DG. Electrocardiographic Biomarkers for Detection of Drug-Induced Late Sodium Current Block. PLoS One. 2016 Dec 30;11(12):e0163619. doi: 10.1371/journal.pone.0163619. eCollection 2016. PMID 28036334
- [Derived] Johannesen L, Vicente J, Hosseini M, Strauss DG. Automated Algorithm for J-Tpeak and Tpeak-Tend Assessment of Drug-Induced Proarrhythmia Risk. PLoS One. 2016 Dec 30;11(12):e0166925. doi: 10.1371/journal.pone.0166925. eCollection 2016. PMID 28036330
- Available data/document: ECG, PK and clinical information database: doi:10.13026/C2HP45 — https://physionet.org/physiobank/database/ecgrdvq/ — This publicly available database contains raw and annotated ECG signals, PK measures as well as clinical information of this study.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 healthy volunteers were assessed for eligibility. 24 subjects were excluded because they did not meet the inclusion criteria. 22 of 28 subjects who met the inclusion criteria were randomized and allocated to receive crossed-over intervention. Williams Latin square design balanced for first-order carryover effects was used for randomization.
Groups:
- Ranolazine 1500 mg: Single oral dose of Ranolazine 1500mg. Each subject received each drug only once in a randomized sequence (10 sequences in total).
- Dofetilide 500 mcg: Single oral dose of Dofetilide 500mcg. Each subject received each drug only once in a randomized sequence (10 sequences in total).
- Verapamil HCl 120 mg: Single oral dose of Verapamil HCl 120 mg. Each subject received each drug only once in a randomized sequence (10 sequences in total).
- Quinidine Sulfate 400 mg: Single oral dose of Quinidine sulfate 400mg. Each subject received each drug only once in a randomized sequence (10 sequences in total).
- Placebo: Single oral dose of Placebo (comparison group). Each subject received each drug only once in a randomized sequence (10 sequences in total).
Period: Period 1
Arm/Group | Ranolazine 1500 mg | Dofetilide 500 mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400 mg | Placebo
Started | 5 | 4 | 5 | 4 | 4
Completed | 5 | 4 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Ranolazine 1500 mg | Dofetilide 500 mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400 mg | Placebo
Started | 5 | 4 | 4 | 4 | 5
Completed | 5 | 4 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Ranolazine 1500 mg | Dofetilide 500 mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400 mg | Placebo
Started | 4 | 4 | 5 | 5 | 4
Completed | 4 | 4 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Ranolazine 1500 mg | Dofetilide 500 mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400 mg | Placebo
Started | 4 | 5 | 4 | 4 | 5
Completed | 4 | 5 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Ranolazine 1500 mg | Dofetilide 500 mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400 mg | Placebo
Started | 4 | 5 | 4 | 4 | 4
Completed | 4 | 5 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either ranolazine, dofetilide, verapamil, quinidine or placebo.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White / Not Hispanic or Latino | 16
  White / Hispanic or Latino | 1
  African American / Not Hispanic or Latino | 4
  Asian / Not Hispanic or Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 22
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (2.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 107.1 (8.5)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 59.7 (7.2)
Heart rate [Mean (Standard Deviation); unit: beats per minute (bpm)] | 56.8 (6.4)
PR interval [Mean (Standard Deviation); unit: ms] | 162.1 (21.6)
QRS duration [Mean (Standard Deviation); unit: ms] | 97.4 (6.7)
J-Tpeakc (heart rate corrected J-Tpeak interval) [Mean (Standard Deviation); unit: ms] | 225.6 (19.8)
Tpeak-Tend interval [Mean (Standard Deviation); unit: ms] | 73.1 (6.4)
QTc (Fridericia's heart rate corrected QT interval) [Mean (Standard Deviation); unit: ms] | 395.9 (17.1)
Spatial QRS-T angle [Mean (Standard Deviation); unit: degrees] | 34.5 (9.9)
Ventricular gradient [Mean (Standard Deviation); unit: mV*ms] | 111.4 (29.5)

OUTCOME MEASURES:

1. Primary Outcome: Placebo, and Baseline-adjusted Changes in PR, QRS, J-Tpeak, Tpeak-Tend and QTc
Description: Compute maximum mean placebo, and baseline-adjusted change for: PR (ms), QRS (ms), J-Tpeak (ms), Tpeak-Tend (ms) and QTc (ms)
Time Frame: 24 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: ms
Groups:
- Ranolazine 1500mg: Single oral dose of Ranolazine 1500mg
- Dofetilide 500mcg: Single oral dose of Dofetilide 500mcg
- Verapamil HCl 120 mg: Single oral dose of Verapamil HCl 120 mg
- Quinidine Sulfate 400mg: Single oral dose of Quinidine sulfate 400mg
Arm/Group | Ranolazine 1500mg | Dofetilide 500mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 22 | 22 | 21
ms
  Change in PR interval | 6.5 [1.1 to 11.8] | 2.3 [-3.0 to 7.6] | 32.1 [26.7 to 37.4] | 5.1 [-0.3 to 10.5]
  Change in QRS duration | 2.7 [0.5 to 4.9] | 1.1 [-1.1 to 3.3] | 2.6 [0.4 to 4.8] | 2.1 [-0.2 to 4.3]
  Change in J-Tpeakc | 3.3 [-3.4 to 9.9] | 39.5 [32.8 to 46.2] | -2.4 [-9.0 to 4.3] | 29.1 [22.4 to 35.9]
  Change in Tpeak-Tend | 8.8 [1.9 to 15.8] | 40.0 [33.0 to 46.9] | 4.8 [-2.2 to 11.7] | 49.8 [42.8 to 56.8]
  Change in QTc | 12.6 [5.5 to 19.6] | 79.3 [72.2 to 86.3] | 5.2 [-1.8 to 12.2] | 78.1 [70.9 to 85.2]
Statistical Analysis 1: Comparison: Ranolazine 1500mg vs Dofetilide 500mcg vs Verapamil HCl 120 mg vs Quinidine Sulfate 400mg; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — For each ECG biomarker and treatment, the null hypothesis is that there is no difference in the biomarker change from baseline between the treatment and placebo; For each ECG biomarker and treatment, the placebo-corrected change from baseline was computed using linear mixed effect model

2. Primary Outcome: Placebo, and Baseline-adjusted Changes in Spatial QRS-T Angle
Description: Compute maximum mean placebo, and baseline-adjusted change for: spatial QRS-T angle (degrees)
Time Frame: 24 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Ranolazine 1500mg | Dofetilide 500mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 22 | 22 | 21
degrees | -2.2 [-4.6 to 0.1] | -4.9 [-7.2 to -2.6] | -2.4 [-4.4 to 0.3] | 3.9 [1.6 to 6.3]
Statistical Analysis 1: Comparison: Ranolazine 1500mg vs Dofetilide 500mcg vs Verapamil HCl 120 mg vs Quinidine Sulfate 400mg; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Placebo, and Baseline-adjusted Changes in Ventricular Gradient
Description: Compute maximum mean placebo, and baseline-adjusted change for: ventricular gradient (mV*ms).
Time Frame: 24 hours
Measure: Least Squares Mean (95% Confidence Interval); unit: mV*ms
Arm/Group | Ranolazine 1500mg | Dofetilide 500mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 22 | 22 | 21
mV*ms | 2.5 [-1.8 to 6.8] | 4.8 [0.5 to 9.1] | 4.2 [-0.1 to 8.5] | 6.0 [1.6 to 10.3]
Statistical Analysis 1: Comparison: Ranolazine 1500mg vs Dofetilide 500mcg vs Verapamil HCl 120 mg vs Quinidine Sulfate 400mg; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Relationship (Ratio) Between Heart Rate and QT
Description: Different post-dose time-points employ different techniques for altering heart rate (leg raises and postural maneuvers). Using the measurements from all the time-points of postural maneuvers, the QT/RR relationship was modeled as a linear relationship between the square root of RR in seconds and QT in seconds and computed on a by subject, treatment and time-point basis. The change in the QT and heart rate relationship was assessed as the difference (mean and 95% CI) between the slopes from the models for each drug vs. placebo.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Ranolazine 1500mg | Dofetilide 500mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 22 | 22 | 21
ratio | 0.01 [-0.02 to 0.05] | 0.06 [0.02 to 0.09] | 0.02 [-0.01 to 0.06] | 0.11 [0.07 to 0.14]

5. Secondary Outcome: Change in PR, QRS, J-Tpeak, Tpeak-Tend and QTc Using Exposure/Response (Dofetilide and Verapamil Arms)
Description: The exposure response analysis will be performed for each treatment and will use a linear or nonlinear model (as determined by visual inspection) to quantify the relationship between exposure and Baseline and placebo adjusted change from Baseline for each ECG parameter (same as for primary analysis).
  The magnitude of change (mean and 95% CI) in QTc for the observed mean Cmax for each drug may be calculated.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: ms per ng/ml
Arm/Group | Dofetilide 500mcg | Verapamil HCl 120 mg
Number analyzed (Participants) | 22 | 22
ms per ng/ml
  Change in PR | -0.5 [-3.2 to 2.2] | 28.7 [22.9 to 34.5]
  Change in QTc | 73.6 [65.8 to 81.5] | 3.9 [-0.7 to 8.5]
  Change in QRS | 0.2 [-1.7 to 2.1] | 0.3 [-1.8 to 2.4]
  Change in J-Tpeakc | 39.1 [31.6 to 46.6] | -0.7 [-4.5 to 3.0]
  Change in Tpeak-Tend | 34.4 [26.9 to 42.0] | 3.6 [1.9 to 5.4]

6. Secondary Outcome: Change in PR, QRS, J-Tpeak, Tpeak-Tend and QTc Using Exposure/Response (Ranolazine and Quinidine Arms)
Description: as for outcome 5
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: ms per mcg/ml
Arm/Group | Ranolazine 1500mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 21
ms per mcg/ml
  Change in PR | 4.2 [0.8 to 7.6] | 3.0 [-0.8 to 6.8]
  Change in QTc | 12.0 [7.3 to 16.7] | 78.9 [68.2 to 89.7]
  Change in QRS | 0.8 [-0.9 to 2.6] | 0.4 [-1.8 to 2.6]
  Change in J-Tpeakc | 0.7 [-3.3 to 4.7] | 26.1 [13.5 to 38.7]
  Change in Tpeak-Tend | 10.0 [7.3 to 12.7] | 51.2 [34.6 to 67.8]

7. Secondary Outcome: Change in Spatial QRS-T Angle Using Exposure/Response (Dofetilide and Verapamil Arms)
Description: The exposure response analysis will be performed for each treatment and will use a linear or nonlinear model (as determined by visual inspection) to quantify the relationship between exposure and Baseline and placebo adjusted change from Baseline for each ECG parameter (same as for primary analysis).
  The magnitude of change (mean and 95% CI) in spatial QRS-T angle for the observed mean Cmax for each drug may be calculated.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: degrees per ng/ml
Arm/Group | Dofetilide 500mcg | Verapamil HCl 120 mg
Number analyzed (Participants) | 22 | 22
degrees per ng/ml | -3.9 [-5.4 to -2.4] | 0.4 [-1.0 to 1.9]

8. Secondary Outcome: Change in Spatial QRS-T Angle Using Exposure/Response (Ranolazine and Quinidine Arms)
Description: as for outcome 7
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: degrees per mcg/ml
Arm/Group | Ranolazine 1500mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 21
degrees per mcg/ml | -1.0 [-2.62 to 0.67] | 2.7 [-0.3 to 5.8]

9. Secondary Outcome: Change in Ventricular Gradient Using Exposure/Response (Dofetilide and Verapamil Arms)
Description: The exposure response analysis will be performed for each treatment and will use a linear or nonlinear model (as determined by visual inspection) to quantify the relationship between exposure and Baseline and placebo adjusted change from Baseline for each ECG parameter (same as for primary analysis).
  The magnitude of change (mean and 95% CI) in ventricular gradient for the observed mean Cmax for each drug may be calculated.
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: mV.ns per ng/ml
Arm/Group | Dofetilide 500mcg | Verapamil HCl 120 mg
Number analyzed (Participants) | 22 | 22
mV.ns per ng/ml | 4.0 [0.6 to 7.5] | 1.2 [-1.5 to 3.4]

10. Secondary Outcome: Change in Ventricular Gradient Using Exposure/Response (Ranolazine and Quinidine Arms)
Description: as for outcome 9
Time Frame: 24 hours
Measure: Mean (95% Confidence Interval); unit: mV.ns per mcg/ml
Arm/Group | Ranolazine 1500mg | Quinidine Sulfate 400mg
Number analyzed (Participants) | 22 | 21
mV.ns per mcg/ml | -0.7 [-3.8 to 2.4] | 1.6 [-2.1 to 5.2]

ADVERSE EVENTS:
Time Frame: From May 2013 to July 2013
Groups:
- Placebo: Single oral dose of Placebo (comparison group)
Arm/Group | Ranolazine 1500mg | Dofetilide 500mcg | Verapamil HCl 120 mg | Quinidine Sulfate 400mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 4/22 | 6/22 | 6/22 | 12/21 | 3/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine 1500mg (N=22) | Dofetilide 500mcg (N=22) | Verapamil HCl 120 mg (N=22) | Quinidine Sulfate 400mg (N=21) | Placebo (N=22)
Dizziness (Nervous system disorders) | 3 (4) | 2 (2) | 4 (4) | 8 (8) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No